CLINICAL TRIAL: NCT06144177
Title: Induction in the Dark: a Prospective Randomized Control Trial for Perioperative Pediatric Anxiety
Brief Title: Induction in the Dark
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Natalie Barnett, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00132312
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Darkened room and star projector with parental presence (Active Comparator): Subjects assigned to this arm, when in the operating room prior to the start of induction, the room will be darkened, and a star projector that lights up the ceiling and walls will be turned on. They will also have a parent in the room with them during induction of anesthesia.
  Interventions: Other: Dark with star projector; Other: Parental Presence
- Preoperative midazolam 0.5 mg/kg po and parental presence (Active Comparator): Subjects assigned to this arm will be given midazolam by mouth preoperatively, and will have a parent in the room with them during induction of anesthesia.
  Interventions: Drug: Preoperative midazolam; Other: Parental Presence
- Parental presence alone (Active Comparator): Subjects assigned to this arm will have a parent in the room with them during induction of anesthesia.
  Interventions: Other: Parental Presence

INTERVENTIONS:
Other: Dark with star projector — When in the operating room prior to the start of induction, the room will be darkened, and a star projector that lights up the ceiling and walls will be turned on.
  Arms: Darkened room and star projector with parental presence
Drug: Preoperative midazolam — Midazolam by mouth preoperatively.
  Arms: Preoperative midazolam 0.5 mg/kg po and parental presence
Other: Parental Presence — A parent or guardian will accompany the child into the OR and be present for the start of induction.

SUMMARY:
This study will enroll children ages 2-6 who are undergoing an elective outpatient surgical procedure under general anesthesia. They will be randomized to one of the following groups and assessed for preoperative anxiety, mask acceptance, and behavioral changes in the following week.

1. darkened room and star projector with parental presence;
2. preoperative midazolam 0.5 mg/kg by mouth and parental presence; or
3. parental presence alone.

ELIGIBILITY:
Inclusion Criteria

* Age 2 to 6 years old
* American Society of Anesthesiologists physical status I-II
* Outpatient elective surgical procedures
* Undergoing general anesthesia
* Parent or guardian willing to be present during induction

Exclusion Criteria

* History of previous surgery
* Fear of the dark
* Contraindication to inhalational mask induction of general anesthesia such as allergy to inhalation medication, NPO violation, active nausea or vomiting, severe GERD, etc.
* Severe developmental delay
* Severe obvious, preoperative anxiety
* Patients currently using psychiatric medications
* Non-English speaking

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Mask acceptance | during induction evaluated up until the start of the scheduled surgery
  Mask acceptance during inhalational mask induction as measured by the mask acceptance scale (MAS). The MAS is scored on a scale from 1-4 by evaluating if the child is calm and accepting of the mask (4), slightly scared but easily calmed (3), has moderate fear of the mask and is not easily calmed (2), or cries, screams, or is terrified (1) during induction when using the inhalation mask. A higher score is better.

SECONDARY OUTCOMES:
Perioperative anxiety | Measured preoperatively, then measured again during the entry to operating room.
  Perioperative anxiety will be measured using the modified Yale perioperative anxiety scale (mYpas) at two different time points; the first will be measured preoperatively in holding, and the other will be measured again during the entry to the operating room. The mYpas consists of 22 items, divided into five categories: activity, vocalizations, emotional expressivity, state of apparent arousal, and use of parent. The evaluator will rate the subject in each category (he highest behavioral level observed in each of the five m-YPAS categories is the score for that category), then divide each item rating by the highest possible rating, add all of the produced values, multiply by 100, then divide by 2. The lower the score, the less anxiety the patient is exhibiting.
Parental satisfaction of induction experience | evaluated after child's induction is complete up until the end of surgery
  After the induction period of anesthesia is over, the parent or guardian who accompanied the child to the operating room and was present for induction will complete a satisfaction survey. There are 6 questions rated from 1-5 (1 being strongly disagree, and 5 being strongly agree) asking how they felt about the induction experience. There is one question asking about how the parent felt about the child's acceptance of the mask during induction. This is rated from 1 (poor) to 4 (excellent). The scores given for each question are added up. Scores can range from 7-29. The higher the score, the better outcome and higher satisfaction.
Post-Operative Emergency Delirium | from PACU arrival until discharge
  Once in the PACU, the patient will be evaluated for emergence delirium using the Pediatric Anesthesia Emergence Delirium (PAED) Scale. The evaluator will answer 3 questions about the patient's actions on a scale from 0 (extremely) to not at all (1), then an additional 2 questions about restlessness and inconsolable, scored from 0 (not at all) to 4 (extremely. The scores are added up. The total score can range from 0-20, and the lower the score, the better.
Behavioral Changes | Day 1 Post-Op and Day 7 Post-Op, up to 30 days post-operatively
  At Day 1 Post-Op and again at Day 7 Post Op, a parent or guardian will answer a series of 27 questions that evaluate the child for behavioral changes occurring post-operatively by using the Post-Hospitalization Behavior Questionnaire (PHBQ). The rating scale for this assessment has 5 response options: (1) less than before (2), same as before (3), more than before (4), and much more than before (5). The answerers are added up with a possible range of 27-135. The lower the score, the less behavioral changes have occurred since the procedure.
Time to PACU discharge | time in recovery, up to 30 days post-op
  The time in recovery will be measured from time in recovery starts, to time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Barnett, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided